CLINICAL TRIAL: NCT03142646
Title: Safety and Efficacy Evaluation of IM19 CAR-T Cells on Refractory or Relapsed B-ALL Patients
Brief Title: Safety and Efficacy Evaluation of IM19 CAR-T Cells
Acronym: IM19CAR-T
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2016-06-06; First posted 2017-05-05 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2017-10

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

ARMS (1):
- IM19 CART (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by a single infusion of IM19CART cells administered intravenously.
  Interventions: Biological: IM19 CAR-T

INTERVENTIONS:
Biological: IM19 CAR-T — All patients will be treated with fludarabine and cyclophosphamide for 3 days,then,CAR-T cells expressing CD19 CAR will be infused 24-96 hours later.
  Other Names: fludarabine，cyclophosphamide

SUMMARY:
Assessment of the Safety and Feasibility of Administering T Cells Expressing an Anti-CD19 Chimeric Antigen Receptor to Patients With CD19+ B-cell leukemia or CD19+ B-all.

DETAILED DESCRIPTION:
Assessment of the Safety and Feasibility of Administering T Cells Expressing an Anti-CD19 Chimeric Antigen Receptor to Patients With CD19+ B-cell leukemia or CD19+ B-ALL patients and determine the MTD,LTD and the best dosage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD19+ leukemia, meeting the following criteria

  * At least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody (Rituximab) therapy)
  * Less than 1 year between last chemotherapy and progression
  * Not eligible or appropriate for allo-HSCT
* To be aged 4 to 65 years
* Estimated survival of ≥ 6 months, but ≤ 2 years
* ECOG score ≤2
* Relapse after auto-HSCT
* Women of childbearing potential must have a urine pregnancy test taken and proven negative prior to the treatment. All patients agree to use reliable methods of contraception during the trial period and until follow-up for the last time.
* Voluntary participation in the clinical trials and sign the informed consent.

Exclusion Criteria:

* History of epilepsy or other CNS disease
* Patients have GVHD, which needs treatment with immunosuppressive agents
* Patients with prolonged QT interval or severe heart disease
* Patients in pregnancy or breast-feeding period
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* Previously treatment with any gene therapy products
* Feasibility assessment during screening demonstrates <30% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation
* ALT /AST>3 x normal value; Creatinine> 2.5 mg/dl; Bilirubin >2.0 mg/dl
* Any uncontrolled medical disorders that the researchers consider are not eligible to participate the clinical trial
* HIV infection
* Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08-30 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 2 years
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria 2.

SECONDARY OUTCOMES:
Overall response rate | 2 years
  An objective response is defined as: (1) a morphologic complete response (CR) or (2) a complete response with incomplete recovery of counts (CRi) (based on NCCN guidelines (National Comprehensive Cancer Network (NCCN), 2014) or (3) a negative minimal residual disease assessed by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: hui liu, MD, Principal Investigator — Beijing Hospital
Locations (2):
- China (2):
  - Beijing hospital, Beijing
  - Peking University People's Hospital (PKUPH), Beijing

IPD SHARING:
Plan to Share IPD: No